CLINICAL TRIAL: NCT03969615
Title: SuperNO2VA™ and General Anesthesia Postoperative Care: Comparing the Incidence, Severity, and Duration of Postoperative Oxygen Desaturation Between SuperNO2VA™ and Standard of Care, a RCT
Brief Title: SuperNO2VA™ and General Anesthesia Postoperative Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vyaire Medical (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0371
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Hypoxemia; Acute Respiratory Failure
MeSH Terms: conditions — Hypoxia | interventions — Cannula; Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Supplemental oxygen (Active Comparator): 5lpm of supplemental oxygen via a nasal cannula or face mask
  Interventions: Device: Supplemental oxygen
- SuperNO2VA nasal positive airway pressure device (Experimental): Intervention arm will receive the SuperNO2VA nasal positive pressure device at 10lpm
  Interventions: Device: SuperNO2VA nasal positive airway pressure devic

INTERVENTIONS:
Device: SuperNO2VA nasal positive airway pressure devic — SuperNO2VA nasal positive airway pressure device utilizes supplemental oxygen and an adjustable pressure limiting valve to maintain upper airway latency
  Arms: SuperNO2VA nasal positive airway pressure device
Device: Supplemental oxygen — 5lpm of supplemental oxygen
  Other Names: nasal cannula; face mask
  Arms: Supplemental oxygen

SUMMARY:
The purpose of the study is to randomly and prospectively evaluate the differences in outcomes between the control group (closed full facemask immediate post-extubation with standard oxygenating device used post-operatively in PACU) and the SuperNO2VA™ group (SuperNO2VA™ immediate post-extubation and post-operatively in PACU)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older
2. Patients scheduled for general anesthesia with a supraglottic device or ETT
3. American Society of Anesthesiology (ASA) Physical Status I-IV (E)
4. Has provided written informed consent
5. BMI > 35 kg/m2 or documented Obstructive Sleep Apnea

Exclusion Criteria:

1. Inability to give informed consent
2. ASA V (E)
3. Allergy to Propofol
4. Any condition, in the Investigator's opinion, that would conflict or otherwise prevent the subject from complying with study required procedures, schedule or other study conduct
5. BMI < 35 kg/m2 with no documented diagnosis (known) of Obstructive Sleep Apnea
6. Known diagnosis of moderate to severe COPD/lung disease
7. Patients that remained intubated post-operatively
8. Patient refusal to wear the treatment device (SuperNO2VA™, nasal cannula, or oxygen facemask) for the duration of the study period postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-10-15 (Estimated)

PRIMARY OUTCOMES:
Hypoxemia | Within 90 minutes of extubation between the two study groups.
  Compare the incidence, severity, and duration of postoperative oxygen desaturation (oxygen saturation below 90% for greater than 1 consecutive minute)

SECONDARY OUTCOMES:
Airway maneuvers | Within 90 minutes of extubation
  Compare the number of airway interventions including chin up and/or jaw thrust, oral and/or nasal airway insertion, mask ventilation, intubation with ETT or SGA insertion performed by anesthesia providers
Post op respiratory complications | Within 90 minutes of extubation
  Compare the incidence of respiratory complications between the two groups (shortness of breath, respiratory rate > 20 breaths per minute, accessory muscle use, difficulty breathing/swallowing/speaking)
Length of PACU stay | Within 24 hours of surgery
  Compare the length of stay (time ready for discharge) in the recovery period between the control group and the SuperNO2VA™ group.

CONTACTS AND LOCATIONS:
Overall Officials: Carin Hagberg, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas, MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sun Z, Sessler DI, Dalton JE, Devereaux PJ, Shahinyan A, Naylor AJ, Hutcherson MT, Finnegan PS, Tandon V, Darvish-Kazem S, Chugh S, Alzayer H, Kurz A. Postoperative Hypoxemia Is Common and Persistent: A Prospective Blinded Observational Study. Anesth Analg. 2015 Sep;121(3):709-715. doi: 10.1213/ANE.0000000000000836. PMID 26287299
- [Result] Simonneau G, Vivien A, Sartene R, Kunstlinger F, Samii K, Noviant Y, Duroux P. Diaphragm dysfunction induced by upper abdominal surgery. Role of postoperative pain. Am Rev Respir Dis. 1983 Nov;128(5):899-903. doi: 10.1164/arrd.1983.128.5.899. PMID 6638679
- [Result] Mutter TC, Chateau D, Moffatt M, Ramsey C, Roos LL, Kryger M. A matched cohort study of postoperative outcomes in obstructive sleep apnea: could preoperative diagnosis and treatment prevent complications? Anesthesiology. 2014 Oct;121(4):707-18. doi: 10.1097/ALN.0000000000000407. PMID 25247853
- [Result] Abdelsattar ZM, Hendren S, Wong SL, Campbell DA Jr, Ramachandran SK. The Impact of Untreated Obstructive Sleep Apnea on Cardiopulmonary Complications in General and Vascular Surgery: A Cohort Study. Sleep. 2015 Aug 1;38(8):1205-10. doi: 10.5665/sleep.4892. PMID 25761980
- [Result] Smith PL, Wise RA, Gold AR, Schwartz AR, Permutt S. Upper airway pressure-flow relationships in obstructive sleep apnea. J Appl Physiol (1985). 1988 Feb;64(2):789-95. doi: 10.1152/jappl.1988.64.2.789. PMID 3372436
- [Result] Cabrini L, Nobile L, Plumari VP, Landoni G, Borghi G, Mucchetti M, Zangrillo A. Intraoperative prophylactic and therapeutic non-invasive ventilation: a systematic review. Br J Anaesth. 2014 Apr;112(4):638-47. doi: 10.1093/bja/aet465. Epub 2014 Jan 19. PMID 24444661
- [Result] Neligan PJ, Malhotra G, Fraser M, Williams N, Greenblatt EP, Cereda M, Ochroch EA. Continuous positive airway pressure via the Boussignac system immediately after extubation improves lung function in morbidly obese patients with obstructive sleep apnea undergoing laparoscopic bariatric surgery. Anesthesiology. 2009 Apr;110(4):878-84. doi: 10.1097/ALN.0b013e31819b5d8c. PMID 19293693
- [Result] Jaber S, De Jong A, Castagnoli A, Futier E, Chanques G. Non-invasive ventilation after surgery. Ann Fr Anesth Reanim. 2014 Jul-Aug;33(7-8):487-91. doi: 10.1016/j.annfar.2014.07.742. Epub 2014 Aug 29. PMID 25168304